CLINICAL TRIAL: NCT03232749
Title: Predicting Response to Intra-Articular Corticosteroid Injection in Patients With Osteoarthritis of the Glenohumeral Joint
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The physician in charge is leaving the University of Florida
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201700603-A; OCR18320 (Other: University of Florida)
Record Dates: First submitted 2017-06-26; First posted 2017-07-28 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis of the Glenohumeral Joint
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Acetate; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- symptomatic primary osteoarthritis of the shoulder (Other): Subjects enrolled into the study will be those who have failed previous treatment including over-the-counter analgesics and activity modification, and have elected to receive a medically-indicated, ultrasound-guided IACSI in the shoulder
  Interventions: Procedure: intraarticular corticosteroid injections (IACSI); Drug: corticosteroid injections; Device: Ultrasound

INTERVENTIONS:
Procedure: intraarticular corticosteroid injections (IACSI) — ultrasound-guided IACSI will be administered
Drug: corticosteroid injections — Corticosteroid will be administered is used to treat pain and swelling that occurs with arthritis and other joint disorder
  Other Names: Methylprednisolone, Depo-medrol
Device: Ultrasound — ultrasound-guided IACSI

SUMMARY:
This study will examine the effectiveness of a single cortisone injection in patients with shoulder osteoarthritis over a 6-month period, and identify clinical and radiographic factors to help predict how a patient with shoulder osteoarthritis will respond to a cortisone injection utilizing ultrasound guidance.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of intraarticular corticosteroid injections (IACSI) for glenohumeral arthritis by 1) through patient-reported outcomes and 2) identifying clinical and radiographic predictors of IACSI success.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of symptomatic primary osteoarthritis of the shoulder will be recruited from the patient population seeking treatment at the Orthopaedics Sports Medicine Institute.
* those who have failed previous treatment including over-the-counter analgesics and activity modification
* have elected to receive a medically-indicated, ultrasound-guided IACSI in the shoulder.

Exclusion Criteria:

* Patients will be excluded from the study for any of the following reasons:
* Post traumatic osteoarthritis
* Inflammatory osteoarthritis
* Imaging confirmed rotator cuff tear
* Prior ipsilateral shoulder surgery
* Memory loss or inability to complete study measures
* History of allergy to injection medications
* Diabetic patients with patient-reported fasting blood glucose >200
* Prior injection in the ipsilateral shoulder within three months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Schoch, M.D., Principal Investigator — Faculty
Locations (2):
- United States (2):
  - UF and Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida
  - UF Health Orthopaedics and Sports Medicine Institute, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
Started | 25
Completed | 21
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: ASES Scores at Each Time Point
Description: ASES (American Shoulder & Elbow Surgeon) score. Data points a change for all pre-specified time points and is reported. ASES has 11 items scored by Pain VAS (1 question) Function (10 questions); Score: 0-100 (Higher score is better).
Time Frame: Baseline, 2 weeks, 1 month, 2 months, 3 months, 6 months
Population: All participants did not return for all outcome measure time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
Number analyzed (Participants) | 25
score on a scale
  Baseline ASES score | 48.52 (13.18)
  2 Week ASES score | 79.72 (23.32)
  1 Month ASES scrore | 73.86 (28.24)
  2 Month ASES score: number analyzed (Participants) | 22
  2 Month ASES score | 28.60 (28.57)
  3 Month ASES score: number analyzed (Participants) | 22
  3 Month ASES score | 71.78 (22.34)
  6 Month ASES score: number analyzed (Participants) | 16
  6 Month ASES score | 61.48 (25.78)

2. Primary Outcome: Visual Analog Scale Scores at Each Time Point.
Description: VAS (Visual Analog Scale) pain score improvement > 1.4 points (The number that the respondent indicates on the scale to rate their pain intensity is recorded. Scores range from 0=no pain and 10=worst pain). The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0=no pain and 10=worst pain.
Time Frame: Baseline, post-injection (5-10 minutes), 2 weeks, 1 month, 2 months, 3 months, 6 months
Population: All participants did not return for all outcome measure time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
Number analyzed (Participants) | 25
score on a scale
  Baseline VAS score | 4.54 (2.62)
  Post-injection VAS score | 1.86 (1.80)
  2 Weeks VAS score: number analyzed (Participants) | 24
  2 Weeks VAS score | 1.18 (1.59)
  1 Month VAS score | 2.05 (2.06)
  2 Month VAS score: number analyzed (Participants) | 22
  2 Month VAS score | 2.56 (2.97)
  3 Month VAS score: number analyzed (Participants) | 22
  3 Month VAS score | 2.50 (2.38)
  6 Month VAS score: number analyzed (Participants) | 16
  6 Month VAS score | 2.44 (3.05)

3. Primary Outcome: SST (Simple Shoulder Test) Scores at Each Time Point
Description: SST (Simple Shoulder Test) score improvement > 2.4 points. 12 items that are answered yes/no (measures functional limitations of the affected shoulder): Scored: 0-12 (Higher score is better)
Time Frame: Baseline, 2 weeks, 1 month, 2 months, 3 months, 6 months
Population: All participants did not return for all outcome measure time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
Number analyzed (Participants) | 25
score on a scale
  Baseline SST Score | 5.29 (2.46)
  2 Week SST Score: number analyzed (Participants) | 22
  2 Week SST Score | 8.40 (2.36)
  1 Month SST Score: number analyzed (Participants) | 24
  1 Month SST Score | 7.32 (3.82)
  2 Month SST Score: number analyzed (Participants) | 19
  2 Month SST Score | 5.92 (3.43)
  3 Month SST Score: number analyzed (Participants) | 19
  3 Month SST Score | 6.73 (3.32)
  6 Month SST Score: number analyzed (Participants) | 15
  6 Month SST Score | 7.00 (2.73)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Symptomatic Primary Osteoarthritis of the Shoulder
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03232749/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03232749/ICF_001.pdf